CLINICAL TRIAL: NCT00870324
Title: OptiSense Performance in Detecting Atrial Episodes in CRMD Device Patient Population
Brief Title: OptiSense™ Performance in Detecting Atrial Episodes
Acronym: SENSE-AF
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD459
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Tachyarrhythmias; Atrial Fibrillation
Keywords: ICD; Tachyarrhythmias; Atrial Fibrillation; Patients who meets current ICD or CRT-D implant indications
MeSH Terms: conditions — Tachycardia; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1. Control: Patients will receive the Tendril (wide-spaced) lead as part of their ICD implant
  Interventions: Device: Tendril Lead
- 2. Experimental: Patients will receive the OptiSense (narrow-spaced) lead as part of their ICD implant
  Interventions: Device: OptiSense Lead

INTERVENTIONS:
Device: OptiSense Lead — The OptiSense™ Model 1699 lead is a bipolar, steroid-eluting, silicone-insulated, active fixation implantable lead, designed for long-term pacing and sensing in the right atrium. The tip-to-ring spacing in the OptiSense lead is 1.1mm and "narrow-spaced" compared to the Tendril lead.
  Groups: 2. Experimental
Device: Tendril Lead — The Tendril® is a bipolar, steroid-eluting, silicone-insulated, active fixation implantable lead, designed for long-term pacing and sensing in either the atrium or the ventricle. The tip-to-ring spacing in the Tendril is "wide spaced" compared to the OptiSense lead.
  Groups: 1. Control

SUMMARY:
The SENSE-AF study aims to determine the performance of the OptiSense lead in sensing fine episodes of Atrial Tachyarrhythmia/Atrial Fibrillation (AT/AF) and rejecting Far-Field R Wave (FFRW). The performance of the lead will be measured as a difference in device-determined time in AT/AF and surface-ECG determined time in AT/AF. This measurement will be compared to the control group which will be randomized to receive SJM's Tendril™ RA leads.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meets current ICD or CRT-D implant indications and receive a St. Jude Medical ICD/CRT-D
* Patients who will receive a new St. Jude Medical OptiSense or Tendril RA lead as part of their device implant

Exclusion Criteria:

* Patients with a history of Permanent or Persistent AF
* Patient's life expectancy is less than 12 months.
* Patient is pregnant.
* Patient's age at enrollment is less than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with approved pacemaker indications.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the difference in duration between the device-determined time in AF (Device Duration) and the ECG-determined time in AF (ECG Duration). | 3 months post-implant

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - The Ohio State University, Columbus, Ohio